CLINICAL TRIAL: NCT00443339
Title: A Phase II Study of Darbepoetin Alpha in Myelodysplastic Syndromes (MSD)
Brief Title: Darbepoetin Alpha in Myelodysplastic Syndromes (MDS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-DAR500-2006-01
Record Dates: First submitted 2007-03-04; First posted 2007-03-06 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndromes with IPSS Low or Int-1; Anemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Darbepoetin

SUMMARY:
This is an evaluation of the effectiveness of darbepoetin alpha in treating anemia of MDS patients with an International Prognostic Scoring System (IPSS) score of low or intermediate 1.

DETAILED DESCRIPTION:
Inclusion of MDS with IPSS low or int-1 and hemoglobin < 10/dL.

Study drug: Darbepoetin alfa (Aranesp) 500 microg every two weeks subcutaneously during 12 weeks, combined to filgrastim 300 microg twice weekly for an additional 12 weeks in non responders.

Response will be evaluated at 12 weeks. Patients with major or minor erythroid response (HI-E major or minor according to IWG 2000 criteria) will be continued on Aranesp. In non-responders, an additional 12 weeks of Aranesp at the same dosing, combined to Filgrastim (300 ug twice weekly, then adjusted to maintain WBC between 5000 and 10000/mm3) will be proposed. In case of response, the treatment will be continued for a total duration of 24 months. If Hb level reaches levels > 13 g/dl at any time, Aranesp should be discontinued until Hb levels are less than 12 g/dl. Aranesp should then be resumed at 500 µg/injection every 3 weeks. Intervals between injections should be further increased by one week every time they lead to Hb levels > 13 g/dl. The purpose of this dose adjustment is to reach the Aranesp schedule allowing a maintenance Hb level between 11 and 12 g/dl.

ELIGIBILITY:
Inclusion Criteria:

* MDS of the following subtypes:

  * RA, RAS, RAEB with marrow blasts < 10% (according to FAB),
  * RA, RARS, RCMD, RAEB 1, CMML 1 with ≤ 10% WBC counts < 13000/mm3 (according to WHO classification)
* Anemia, defined by Hb < 10 g/dl or RBC transfusion requirement in the absence of other causes of anemia (especially renal failure, iron, or folate deficiency)
* IPSS ≤ 1(ie IPSS low or intermediate 1)
* EPO level < 500 UI/L
* Ability to perform physical tests of exercise tolerance
* No renal failure (creatinine ≤ 120% normal upper value for the center)
* No underlying severe condition
* ECOG performance status score of 0, 1, or 2
* Must be 18 years of age or older at the time of screening
* Written informed consent

Exclusion Criteria:

* Therapy related MDS
* MDS with IPSS > 1 (int 2 or high score)
* Chronic myelomonocytic leukemia with > 10% marrow blasts or WBC > 13000/mm3
* Uncontrolled systemic hypertension
* Cardiac condition: uncontrolled angina, congestive heart failure, or uncontrolled cardiac arrhythmia
* Creatinine level > 120% upper normal value for the center.
* Clinically significant systemic infection or chronic inflammatory disease (eg, rheumatoid arthritis) present at the time of screening
* Serum folate ≤ 2.0 ng/mL or vitamin B12 ≤ 200 pg/mL (anemia related to nutritional deficiencies)
* Other causes of anemia (eg, hemolysis, bleeding, sickle cell anemia, renal disease)
* Pregnant (ie, positive βhCG test) or breast feeding female subjects
* Women of childbearing potential and not using adequate contraceptives
* Known positive antibody response to an erythropoietic growth factor
* Known hypersensitivity to darbepoetin alpha or any of its excipients, or to recombinant erythropoietins
* Patient unable to understand the protocol or to be adequately followed up.
* History of seizures
* Previous history of thrombotic events
* Concomitant treatment with thalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2006-12; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Erythroid response at 12 weeks according to IWG 2000 (major and minor hematologic improvement) and IWG 2006 criteria

SECONDARY OUTCOMES:
Tolerability and safety of darbepoetin alpha
Rate of progression to more severe MDS, with higher IPSS (int 2 or high), or to AML during the treatment and follow-up periods
Overall survival
Quality of life during the study, using the FACT-An and SF36 questionnaires by comparison to pre-treatment values
Overall physical performance as measured by VO2max, 6 minute walk test and the "short physical performance battery" test

CONTACTS AND LOCATIONS:
Overall Officials: Charikleia KELAIDI, MD, Principal Investigator — Groupe Francophone des Myelodysplasies
Locations (28):
- France (28):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU d'Avignon, Avignon
  - CH de la Cote Basque, Bayonne
  - CHU de Brest - Hopital Morvan, Brest
  - CHU de Caen, Caen
  - Hopital Percy, Clamart
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU Albert Michallon, Grenoble
  - CHRU Hurriez, Lille
  - CHRU Limoges, Limoges
  - Hopital Edouard Herriot, Lyon
  - Hopital Paoli Calmette, Marseille
  - Hopital Hotel Dieu, Nantes
  - CHU Archet, Nice
  - Hopital Hotel Dieu, Paris
  - Hopital St Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Jean-Bernard, Poitiers
  - CHU Robert Debre, Reims
  - CHU Pontchaillou, Rennes
  - Hopital Henri Becquerel, Rouen
  - Hopital Hautepierre, Strasbourg
  - Hopital Purpan, Toulouse
  - Hopital Bretonneau, Tours
  - CHU Nancy-Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Kelaidi C, Beyne-Rauzy O, Braun T, Sapena R, Cougoul P, Ades L, Pillard F, Lamberto C, Charniot JC, Guerci A, Choufi B, Stamatoullas A, Slama B, De Renzis B, Ame S, Damaj G, Boyer F, Chaury MP, Legros L, Cheze S, Testu A, Gyan E, Bene MC, Rose C, Dreyfus F, Fenaux P. High response rate and improved exercise capacity and quality of life with a new regimen of darbepoetin alfa with or without filgrastim in lower-risk myelodysplastic syndromes: a phase II study by the GFM. Ann Hematol. 2013 May;92(5):621-31. doi: 10.1007/s00277-013-1686-4. Epub 2013 Jan 29. PMID 23358617